CLINICAL TRIAL: NCT04235075
Title: Computer-assisted Fetal Monitoring - Cardiology
Acronym: SURFAO-CARDIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); University Grenoble Alps (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC19.309
Record Dates: First submitted 2020-01-07; First posted 2020-01-21 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy
Keywords: Signal Database; Pregnancy; Electrocardiogram; Usability; Multimodal signal acquisition

STUDY DESIGN:
Intervention Model Description: Creation of a multimodal database
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnancy volunteer subjects (Experimental): Subjects who will agree to participate in the study will be pregnant women referred to the Grenoble Alpes University Hospital for expert fetal cardiac ultrasound examination who have not revealed any abnormalities.
  Interventions: Device: ECG/PCG and ultrasound signal acquisition

INTERVENTIONS:
Device: ECG/PCG and ultrasound signal acquisition — The ECG - PCG signals are acquired over a 20-minute monitoring phase with passive non invasive sensors (abdominal and thoracic). The volunteer's abdomen is photographed when the electrodes and sensors are installed. An ultrasonography is also performed for 10 minutes.
  The session is filmed for 5 volunteers accepting the video. Any distinctive elements will be removed from photos and videos to prevent the identification of participants.

SUMMARY:
In the context of fetal heart monitoring (prenatal and during childbirth), the SurFAO project offers an alternative to current clinical routines. The challenge is to extract, from non-invasive sensors on the maternal abdomen, a fetal electrocardiogram (ECGf) of great quality allowing a clinical diagnosis (follow-up of the FHR (Fetal Heart Rate)) and extraction of ECG waveforms).

The approach proposes a technological breakthrough shared by a consortium of researchers and clinicians. The originality is driven by innovative methodological choices: the use of a multimodal system (ECG coupling with PCG (phonocardiography)) for the signal acquisition in order to increase the robustness of information extraction, by taking into account clinical uses and the need to support the monitoring process, and by setting up a multimodal database.

The objective is to feed a database that will be used in the future to develop ECGf extraction methods.

DETAILED DESCRIPTION:
To monitor the well-being of a fetus or for clinical diagnosis, the challenge is to extract a high-quality fetal electrocardiogram (fECG) signal from non-invasive sensors on the maternal abdomen.

As early as the 20th week of amenorrhea, heart rhythm disorders (tachycardia, bradycardia) can be detected in the fetus, most often by fortuitous circumstance, during routine obstetrical ultrasound examinations. It is then necessary to analyze these rhythmic anomalies, understand their origin and, if necessary, initiate pharmacotherapy. The effectiveness of the treatments is then monitored by ultrasound in the high-risk pregnancy department.

The analysis of a fetal electrocardiogram (fECG) provides information that allows to determine the nature of the rhythm disorder, its origin and therefore its potential severity.

The innovative methodological approach considered for the extraction of non-invasive ECGf is to combine 2 complementary modalities of the same cardiac phenomenon. This is achieved by combining the use of ECG sensors with sound sensors giving access to phonocardiographic signals (PCG).

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* between 20 and 26 weeks of amenorrhea
* with a BMI between 18.5 and 30 at the beginning of pregnancy
* fetal heart considered normal after expert ultrasound
* examination conditions deemed correct by the expert
* registered in a social security scheme
* having signed the study consent form

Exclusion Criteria:

* subject to a legal protection measure or unable to express consent (guardianship, guardianship) (article L1121-8)
* deprived of liberty by judicial or administrative decision (article L1121-6)
* in a period of exclusion from another study
* with toxic consumption (i.e. tobacco, alcohol, cannabis)
* Intrauterine growth retardation (estimated fetal weight less than the 10th percentile)
* fetal heart rhythm disorders
* with unclear pregnancy term
* with pregnancy denial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
ECG / PCG Signals database | 20 minutes
  Synchronized signals from ECG electrodes and PCG sensors. Signals will be processed to extract fetal ECG and specific waveforms characteristics of fECG (in parts of R waves, P waves, QT intervals, ST intervals).
Ultrasound signals database | 10 minutes
  The fetal heart activity is analyzed using mechanograms and Doppler during ultrasound (gold standard).

SECONDARY OUTCOMES:
Subject acceptability : Score | 10 minutes
  The subject acceptability score will be composed by the addition of 7 scales. These scales have been specifically created for the SurFAO system. The score can go from 0 (worst) to 70 (best). Each scale can give from 0 to 10 points to the final score.
Subject Acceptability : Descriptive analysis | 10 minutes
  Open questions will be asked to the subjects in a questionnaire. A descriptive analysis will be done with the answers.
Use Error evaluation : System Usability Scale (SUS) | 10 minutes
  The System Usability Scale (SUS) is a validated tool for assessing the subjective usability of a system, in this case, the SurFAO System. It contains 10 questions that are rated on a scale from 1 to 5. "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100." Jeff Sauro established the average score of SUS is 68.
  The score can go from 0 (worst) to 100 (best).
Use Error evaluation : Descriptive analysis | 60 minutes
  Difficulties in using the system will be recorded in the case report form and identified using photographs and video. A descriptive analysis will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias LACHUAD, MD, Principal Investigator — University Hospital Grenoble Alpes
Locations (1):
- University Hospital Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noorzadeh S, Rivet B, Gumery PY. An application of Gaussian processes on ocular artifact removal from EEG. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:554-7. doi: 10.1109/EMBC.2015.7318422. PMID 26736322
- [Background] Noorzadeh S, Niknazar M, Rivet B, Fontecave-Jallon J, Gumery PY, Jutten C. Modeling quasi-periodic signals by a non-parametric model: application on fetal ECG extraction. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1889-92. doi: 10.1109/EMBC.2014.6943979. PMID 25570347
- See also: Website of the Clinical Investigation Centre for Innovative Technology of the Grenoble Alpes University Hospital — https://www.cic-it-grenoble.fr/projets/